CLINICAL TRIAL: NCT03161301
Title: Role of IL-37 Genetic Variants in Modulating Innate Immune Response to Periodontal Pathogens
Acronym: ITS
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-0335; R01DE023836 (NIH)
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva, subgingival dental plaque, gingival cervicular fluid and interdental gingival biopsy tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: IL-37 genotype 1.1
- Group 2: IL-37 genotype 1.2
- Group 3: IL-37 genotype 2.2

SUMMARY:
This study will provide mechanistic insight into the underlying causes and molecular level pathogenesis of periodontal diseases. We will identify key mechanisms that confer risk and protection. Ultimately this will lead to new and improved diagnostics and therapeutics. Because periodontal disease is a uniquely accessible biofilm-associated disease it will provide insight into many other diseases such as inflammatory bowel disease and chronic infections associated with indwelling catheters and artificial prostheses. Subjects with periodontal conditions will have therapeutic benefit from the treatments provided.

DETAILED DESCRIPTION:
A maximum of 440 subjects will be enrolled in this study with the goal of identifying 31 of each of the three types of IL-37 genotypes (93 total). Subject participation may include 1 to 9 visits lasting over a period of 6 months. Clinical data and medical history data will be collected at the screening visit to ascertain eligibility. Saliva collected at screening will be used to determine genotype. If one of the three targeted genotypes results, these patients will be assigned to the appropriate genotype group until 31 subjects are in each group at which point recruitment and screening will stop. There are no plans to share genotype classification with subjects. All subjects will have saliva and dental plaque collected at baseline. Twenty four of the 93 subjects (8 from each group) will be selected for gingival biopsy. These 24 subjects will have GCF samples collected at baseline. All subjects will have GCF samples collected at visit 3. Enrolled subjects (31 of each type of the three genotypes) will be recalled up to four additional times spread over twelve weeks for blood collection, to be used for monocyte isolation and whole blood stimulation. Gingival tissue samples will be used for immunohistochemistry, laser capture and RNA extraction. Medical histories, demographics, height and weight, clinical and biological data described above will be recorded and stored on a secure server located at the University of North Carolina. Each participant enrolled into the study will have a unique identification number that has been stripped of any information that could be used by non-study members to identify the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have read, understood and signed an informed consent form in English.
* Subjects must be able and willing to follow study procedures and instructions in English.
* Subjects must be adult Caucasian males or females between the ages of 18 and 65 years (inclusive).
* Subjects must present with at least 20 teeth in the functional dentition, excluding third molars.
* Subjects must have at least 3 teeth in each posterior sextant.

Exclusion Criteria:

* Chronic disease with oral manifestations including diabetes mellitus.
* Current smoker or one that has stopped smoking less than 2 years prior to enrollment.
* Gross oral pathology other than the periodontal disease.
* Treatment with antibiotics for any medical or dental condition within 1 month prior to the screening examination.
* Chronic treatment (i.e., two weeks or more) with any medication known to affect periodontal status (e.g., phenytoin, calcium antagonists, cyclosporin, coumadin, non-steroidal anti-inflammatory drugs, aspirin) within one month of the screening examination.
* Ongoing medications initiated less than three months prior to enrollment (i.e., medications for chronic medical conditions must be initiated at least three months prior to enrollment).
* Significant organ disease including impaired renal function, heart murmur, history of rheumatic fever or valvular disease, or any bleeding disorder.
* Infectious diseases such as hepatitis, HIV or tuberculosis.
* Anemia or other blood dyscrasias.
* Anticoagulant therapy or drugs, such as heparin or warfarin.
* Severe unrestored caries, or any condition that is likely to require antibiotic treatment over the trial.
* Pregnant, or expect to become pregnant within the next several months.
* Females of child-bearing capacity must be willing to have pregnancy test to confirm they are not pregnant.
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult Caucasian male and female subjects recruited from the patients, students and staff at the University of North Carolina at Chapel Hill, as well as the general population in or near Chapel Hill NC.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Cytokines | 6 weeks
  Levels of key cytokines in gingival crevicular fluid.
Gingival Tissue Expression | Baseline
  Levels of IL-37 expressed in gingival tissue samples obtained during routine periodontal treatments.(Immunohistological)
Whole Blood and Monocyte Cytokines | 6 weeks
  Evaluation of cytokine levels in LPS stimulated whole blood and monocytes
mRNA splice variants | Baseline
  Alternate IL-37 mRNA splice variants of gingival tissue among 1.1, 1.2, and 2.2

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Barros, DDS PhD MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No